CLINICAL TRIAL: NCT00959543
Title: MRI Findings in Throwing Shoulders of Waterpolo Players Abnormalities in Professional Waterpolo Players
Brief Title: MRI Findings in Throwing Shoulders of Waterpolo Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Michael A. Badulescu, MD, Kantonal Hospital St. Gallen, Department of Orthopedic Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EKSG09/068
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-06

CONDITIONS: Waterpolo Players; Non Throwing Shoulders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- waterpolo players (Other): 30 throwing shoulders of waterpolo players
  Interventions: Other: MRI
- controle group (Other): 15 healthy patients (non waterpolo players); 30 shoulders
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI and clinical investigation

SUMMARY:
MRI examination of 60 shoulders of waterpolo players (30 throwing shoulders as well as the opposite side) and 15 healthy probands as control group (30 shoulders of non waterpolo players. The correlation of MRI alteration and clinical symptomatic findings in both groups will be investigated. The clinical examination is performed by 2 board certified orthopedic surgeons and based on the Constant Murley Score.

ELIGIBILITY:
Inclusion Criteria:

* Study shoulders of elite waterpolo players
* Study shoulders of healthy non throwing persons
* Age between 18-35 years
* Male
* Given informed consent

Exclusion Criteria:

* Previous shoulder surgery
* Goal keeper
* Metallic implants
* Pacemaker
* Tattoos with metallic colors

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Correlation between alterations of SSP-tendon in MRI and clinical symptoms | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Badulescu, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Department of Orthopedic Surgery, Sankt Gallen, Switzerland